CLINICAL TRIAL: NCT00190164
Title: Evaluation of the Success Rate of a Procedure Without Strict Positioning Post Surgical Versus With Positioning Face Towards the Strict Ground, at Patients Presenting a Macular Hole. Study of Non-Inferiority.
Brief Title: Alleviated Positioning for Small Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P031004; CRC03140
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Macular Hole
Keywords: Macular hole; Vitrectomy; positioning; retina; surgery
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Macular hole surgery with alleviated positioning
  Interventions: Procedure: Macular hole surgery with alleviated positioning
- 2 (No Intervention): Macular hole surgery with no alleviated positioning
  Interventions: Procedure: Macular hole surgery with no alleviated positioning

INTERVENTIONS:
Procedure: Macular hole surgery with alleviated positioning — Macular hole surgery with alleviated positioning
  Arms: 1
Procedure: Macular hole surgery with no alleviated positioning — Macular hole surgery with no alleviated positioning
  Arms: 2

SUMMARY:
Rational of the study: There are arguments to think that the closure of macular holes can be obtained without a strict positioning under certain conditions, i.e. hole size ≤ 400 µm, if the patient avoids the position laid down on the back. In order to be able to confirm these observations, it is necessary to make a randomized study with an adequate number of patients.

Aim of the study: To show that the percentage of success (anatomical closure confirmed by OCT) is not lower in the group without positioning.

Tested Hypothesis: The absence of strict positioning is "at least as effective" on the success of the surgery of small macular holes as the imposition of a strict positioning.

Expected results: To show that the success rate of the surgery of the idiopathic macular holes of 400 µm or less is not decreased by the replacement of a strict positioning (face-down 22h/24) by a simple instruction of avoiding the position laid down on the back, thus avoiding the patients this painful part of the treatment and allowing a reduction in the duration of hospitalization and consequently a reduction in the cost of the treatment.

DETAILED DESCRIPTION:
Rational of the study: There are arguments to think that the closure of macular holes can be obtained without a strict positioning under certain conditions, i.e. hole size ≤ 400 µm, if the patient avoids the position laid down on the back. In order to be able to confirm these observations, it is necessary to make a randomized study with an adequate number of patients.

Main Aim of the study: To show that the percentage of success (anatomical closure confirmed by OCT) is not lower in the group without positioning.

Tested Hypothesis: The absence of strict positioning is "at least as effective" on the success of the surgery of small macular holes as the imposition of a strict positioning.

Primary outcome: Frequency of the successes defined by anatomical closing.

Secondary objectives: To show the non inferiority of the technique without positioning by the following variables: - ETDRS visual acuity in the third postoperative month. - Progression of cataract - Frequency of the complications.

Design of the study: Randomized multicentric study, in parallel groups, open, with individual benefit for the patient.

Number of subjects and duration of the study: 68 patients, divided into two parallel groups, of more than 18 years, presenting a hole ≤ 400 µm, will be included and followed over a period of 3 months. The estimated total duration of the study is 27 months.

Data analysis: In the case of this equivalence clinical trial the margin of non inferiority was fixed at 15%. The secondary criteria will consequently be analyzed.

Expected results: To show that the success rate of the surgery of the idiopathic macular holes of 400 µm or less is not decreased by the replacement of a strict positioning (face-down 22h/24) by a simple instruction of avoiding the position laid down on the back, thus avoiding the patients this painful part of the treatment and allowing a reduction in the duration of hospitalization and consequently a reduction in the cost of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient presenting an idiopathic macular hole of stage 2, 3 or 4
* Opening diameter of the macular hole ≤ 400 µm
* Patient having been informed of the objectives and constraints of the study and having signed an informed consent
* Patient not presenting a per-operational complication having required a complementary gesture or a modification of the usual procedure, with the only exception of discovering a retinal tear, flat, located between 10 and 2h and having required only a treatment by cryo.

Exclusion Criteria:

* Patient having a strong myopia of the eye operated (correction carried or optimal > 6 dioptres)
* Patient MONOPHTALMIA
* Patient presenting a non contact plan capsular CRYSTALLINE being able to leave a passage of gas towards the former segment
* Patient presenting an associated ocular pathology -
* Patient presenting a TM already operated of the eye to include (repetition or failure after a first surgery)
* Patient refusing to sign an assent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Frequency of the successes defined by anatomical closure at third postoperative month. | during the 3 months

SECONDARY OUTCOMES:
Gain of ETDRS visual acuity in the third postoperative month. | during the 3 months
Progression of cataract | during the 7 months
Frequency of the complications | during the 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramin TADAYONI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Ophtalmolgie de l'Hôpital Lariboisière, Paris, France